CLINICAL TRIAL: NCT06461182
Title: Ga-68-CXCR4 PET/CT in Detecting, Evaluating Response to Treatment, and Monitoring Risk of Aggressiveness of Indolent B-cell Lymphoma
Brief Title: Ga-68-CXCR4 PET/CT in Indolent B-cell Lymphoma
Acronym: PentixaFor
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Koo Foundation Sun Yat-Sen Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KF-CXCR4-001
Record Dates: First submitted 2024-05-23; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Indolent B-Cell Non-Hodgkin Lymphoma
Keywords: Ga-68-CXCR4 PET/CT; indolent B-cell lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ga-68-CXCR4 PET/CT in Indolent B-cell Lymphoma (Experimental): Indolent B-cell Lymphoma such as marginal-zone B-cell lymphoma、Waldenstrom macroglobulinemia lymphocytic lymphoma、CLL/SLL、mantle cell lymphoma.
  Interventions: Drug: Ga-68-CXCR4

INTERVENTIONS:
Drug: Ga-68-CXCR4 — Ga-68-CXCR4 for PET/CT procedure in Indolent B-cell Lymphoma
  Other Names: PET/CT

SUMMARY:
This study explores the efficacy of Ga-68-PentixaFor PET/CT in detecting, assessing treatment response, and monitoring the risk of aggressiveness in indolent B-cell lymphoma. The background introduces CXCR4 and discusses its role in cancer research. Currently, FDG-PET is the primary imaging tool for lymphoma staging, but it lacks diagnostic accuracy for low-grade lymphomas. Ga-68-PentixaFor PET demonstrates promising detection capabilities across various lymphomas, suggesting its potential as a superior imaging modality for low-grade lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* The pathological diagnosis is slow-growing lymphoma, such as: marginal-zone B-cell lymphoma, Waldenstrom macroglobulinemia lymphocytic lymphoma, CLL/SLL, mantle cell lymphoma.
* Have undergone or planned to undergo FDG PET scan for indications including initial staging, therapeutic response evaluation, or follow-up examinations within 3 to 6 months in the clinical observation group.
* Able to lie flat for at least 30 minutes.
* Signing the subject consent form.
* ECOG grade 0-2.
* The timing of F-18-FDG usage in this trial follows the "Lymphoma Treatment Principles" of our institution.

Exclusion Criteria:

* Pregnant woman
* Severe renal impairment (eGRF< 30ml/min)
* Known or suspected allergy to radiopharmaceuticals
* Concurrent or previous diagnosis of malignancies other than lymphoma
* Inability to undergo the necessary PET scan procedure
* Refusal or unwillingness to sign the informed consent form
* Severe medical conditions (severe disabilities, mental disorders)

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-04-29 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Performance of Ga-68-CXCR4 PET/CT in indolent B cell lymphoma | up to 24 months
  Detection rate = number of positive scan / total number of scan Sensitivity = number of true positive scan / total number of proven recurrent patient Specificity = number of true negative scan / total number of proven free of disease patient Accuracy = number of (true positive scan + true negative scan) / total number of scan Positive predictive value = number of true positive scan / number of positive scan Negative predictive value = number of true negative scan / number of negative scan

SECONDARY OUTCOMES:
Ga-68-CXCR4 compared to F-18-FDG PET/CT | up to 24 months
  McNemar test, Two-tailed，P<.05
Clinical impact of Ga-68-CXCR4 compared to F-18-FDG PET/CT | up to 24 months
  Treatment plan questionnaires before and after Ga-68-CXCR4 PET/CT
Prognostic value of Ga-68-CXCR4 PET/CT scan | up to 36 months
  The correlation between the radiomic features of Ga-68-CXCR4 PET/CT scan and progression free survival.
  CXCR4 radiomics : Feature extraction was performed with the open-source Python package pyradiomics. For each volume of interest (VOI), including first-order statistics, shape features, grey level co-occurrence matrix (GLCM), grey level run length matrix (GLRLM), grey level size-zone matrix (GLSZM), neighborhood grey level different matrix (NGLDM), and grey level dependence matrix (GLDM).

CONTACTS AND LOCATIONS:
Locations (1):
- Koo Foundation Sun Yat-Sen Cancer Center, Taipei, Beitou, Taiwan